CLINICAL TRIAL: NCT02484833
Title: Erbitux MEtastatic Colorectal Cancer Strategy Study (ERMES): A Phase III Randomized Two Arm Study With FOLFIRI + Cetuximab Until Disease Progression Compared to FOLFIRI + Cetuximab for 8 Cycles Followed by Cetuximab Alone Until Disease Progression in First Line Treatment of Patients With RAS and BRAF Wild Type Metastatic Colorectal Cancer
Brief Title: Erbitux MEtastatic Colorectal Cancer Strategy Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Armando Orlandi (Other)
Responsible Party: Sponsor-Investigator, Armando Orlandi, MD, Ph.D, Catholic University of the Sacred Heart
Organization: Catholic University of the Sacred Heart (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-004299-41
Record Dates: First submitted 2015-04-26; First posted 2015-06-30 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Antineoplastic Agents
Keywords: First line; metastatic colorectal cancer; Cetuximab; strategy study
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOLFIRI + Cetuximab until disease progression (Active Comparator): FOLFIRI + Cetuximab until disease progression
  Interventions: Drug: Cetuximab; Drug: FOLFIRI
- FOLFIRI + Cetuximab followed by Cetuximab alone (Experimental): FOLFIRI + Cetuximab for 8 cycles followed by Cetuximab alone until disease progression
  Interventions: Drug: Cetuximab; Drug: FOLFIRI

INTERVENTIONS:
Drug: Cetuximab
Drug: FOLFIRI

SUMMARY:
* To investigate whether cetuximab alone (given until progression or cumulative toxicity) after 8 cycles of FOLFIRI + cetuximab results in a non inferior Progression Free Survival when compared with continuous FOLFIRI + cetuximab (given until progression or cumulative toxicity).
* To assess whether an improvement in the incidence of grade 3-4 hematological and non-hematological adverse events (AEs) can be achieved in the experimental arm (cetuximab alone after 8 cycles FOLFIRI + cetuximab) as compared to the continuous chemotherapy arm (FOLFIRI plus cetuximab)
* To explore the possibility of using liquid biopsies for molecular profiling as well as monitoring treatment activity in mCRC pts receiving cetuximab based therapy

DETAILED DESCRIPTION:
Survival of patients undergoing therapy with FOLFIRI + cetuximab seems to be related to the ability of this treatment to induce a rapid reduction in tumor mass. In the retrospective analyses of the FIRE-3 trial ETS was significantly associated with PFS and OS, suggesting that ETS reflects the existence of a selected population of patients highly sensitive to cetuximab. This permits the assumption that, once this goal has been achieved, further exposure to combined antineoplastic treatment (cytotoxic drugs and targeted therapy) may not result in improvement or preservation of the result, but only in an increase of side effects that will be additional to unavoidable disease progression. In addition, the heavy exposure to cytotoxic antineoplastic treatments may lead to bone marrow toxicity, hepatic and renal function decreases that could compromise the sequential treatment plan, negatively affecting OS. With the availability of an effective treatment such as cetuximab in monotherapy4 without major side effects on blood counts and liver and kidney function, the use of this treatment alone after achievement of the deepest clinical response could be a viable strategy to achieve a good control of the disease, limiting side effects. As shown in several studies designed to understand the most effective treatment sequence in colorectal carcinoma, the most important factor that influences the overall survival is the possibility to administer more lines of effective therapy. As a consequence, a de-intensifying strategy in a subgroup of highly selected RAS and BRAF WT population might segregate a group of patients with the largest potential for fast-primary treatment. Joining the best induction treatment with the expression of patients capability to undergo additional lines of antineoplastic therapy may be the way to optimize the continuum of care.

Recently, several mechanisms of resistance to anti-EGFR therapy have been described, but until now none may used early in order to support the treatment choice.Moreover, assessment of secondary resistance requires further tissue samples and often it is not really feasible. Therefore, a prospective multiple gene mutation analysis could meet the need of characterizing primary resistance, whereas liquid biopsy might help to recognize resistance occurring early during treatment by means of a simple and repeatable assay. Based on all these considerations, the investigators designed a strategy study: a phase III randomized two arm study with FOLFIRI + cetuximab until disease progression compared to FOLFIRI + cetuximab for 8 cycles followed by cetuximab alone until disease progression in the first line treatment of patients with RAS and BRAF WT metastatic colorectal cancer combined with a prospective multiple gene mutation analysis of both tumor tissue and blood.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of colorectal adenocarcinoma
* Diagnosis of metastatic disease
* RAS and BRAF wildtype
* Measurable disease according to RECIST criteria v1.1
* Male or female over 18 years of age
* ECOG Performance Status 2
* Life expectancy of at least 3 months
* Adequate bone marrow, liver and renal function assessed within 14 days before starting study treatment
* If female and of childbearing potential, have a negative result on a pregnancy test performed a maximum of 7 days before initiation of study treatment
* If female and of childbearing potential, or if male, agreement to use adequate contraception
* Signed informed consent obtained at screening

Exclusion Criteria:

* Any contraindication to use cetuximab, irinotecan, 5 FU or folinic acid
* Active uncontrolled infections or active disseminated intravascular coagulation
* Past or current history of malignancies other than colorectal carcinoma, except for curatively treated basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix
* Pregnancy.
* Breastfeeding.
* Grade III or IV heart failure (NYHA classification)
* Myocardial infarction, unstable angina pectoris, balloon angioplasty (PTCA) with or without stenting within the past 12 months before inclusion in the study
* Cardiac arrhythmias requiring anti-arrhythmic therapy, with the exception of beta blockers or digoxin
* Medical or psychological impairments associated with restricted ability to give consent or not allowing conduct of the study
* Previous chemotherapy for colorectal cancer with the exception of adjuvant treatment, completed at least 6 months before entering the study
* Participation in a clinical study or experimental drug treatment within 30 days prior to study inclusion or during participation in the study
* Known or clinically suspected brain metastases
* History of acute or subacute intestinal occlusion or chronic inflammatory bowel disease or chronic diarrhoea
* Severe, non-healing wounds, ulcers or bone fractures
* Uncontrolled hypertension
* Marked proteinuria (nephrotic syndrome)
* Known DPD deficiency (specific screening not required)
* Known history of alcohol or drug abuse
* A significant concomitant disease which, in the investigating physician's opinion, rules out the patient's participation in the study
* Absent or restricted legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | every 8 weeks from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  PFS
Incidence of grade 3-4 AEs | weekly from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  AEs

SECONDARY OUTCOMES:
Response rate | every 8 weeks from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  RR
Early tumor shrinkage assessed by Response rate at week 8 | at 8 weeks
  ETS
Overall survival | every 8 weeks from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  OS
Cetuximab-related skin toxicity by CTCAE | weekly from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Cetuximab-related skin toxicity
Safety profile assessed by CTCAE | weekly until from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Safety profile
Quality of life assessed by EORT QLQ-C30 and DLQI questionnaires | every 8 weeks from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 32 weeks
  QoL

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy

REFERENCES:
- [Derived] Pinto C, Orlandi A, Normanno N, Maiello E, Calegari MA, Antonuzzo L, Bordonaro R, Zampino MG, Pini S, Bergamo F, Tonini G, Avallone A, Latiano TP, Rosati G, Cogoni AA, Ballestrero A, Zaniboni A, Roselli M, Tamberi S, Barone C. Fluorouracil, Leucovorin, and Irinotecan Plus Cetuximab Versus Cetuximab as Maintenance Therapy in First-Line Therapy for RAS and BRAF Wild-Type Metastatic Colorectal Cancer: Phase III ERMES Study. J Clin Oncol. 2024 Apr 10;42(11):1278-1287. doi: 10.1200/JCO.23.01021. Epub 2024 Jan 5. PMID 38181312